CLINICAL TRIAL: NCT06580340
Title: Effectiveness of an Adapted Physical Activity Program for Subjects Suffering From Haemophilia:a Prospective Interventional Study
Brief Title: Effectiveness of an Adapted Physical Activity Program for Subjects Suffering From Haemophilia
Acronym: EMO-AFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EMO- AFA
Record Dates: First submitted 2024-08-23; First posted 2024-08-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Hemophilia; Sports Physical Therapy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): patients with emophilia receiving a program of adapted physical activity
  Interventions: Other: AFA (Adapted Physical Activity)

INTERVENTIONS:
Other: AFA (Adapted Physical Activity) — An exercise program to improve joint mobility, muscle strength, static and dynamic balance, motor coordination will be performed 2 times/week for 6 months.

SUMMARY:
The present study aims to evaluate the modification of functional capacity induced by an adapted physical activity program in subjects with haemophilia.

The exercise program used aims to improve joint mobility, muscle strength, static and dynamic balance, motor coordination.

The program is structured in 1 hour sessions of 2 days/week and lasts 6 months.

The primary endpoint is the change in functional capacity calculated as the difference between the baseline assessment and the 3 and 6 month assessment of the 6 Minutes Walking Test measured with the G-Walk (BTS Bioengineering S.p.A).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemophilia A or B;
* Signature of informed consent;
* Availability of a medical certificate for non-competitive activities

Exclusion Criteria:

* Active bleeding
* Severe joint deformities that prevent exercise
* Insufficiency of communicative and/or sensory functions so severe that it is impossible to understand or carry out the trainer's instructions (dementia, aphasia, blindness, deafness)
* Heart failure (NYHA class > 2)
* Unstable angina
* Lung disease requiring oxygen therapy
* Symptomatic peripheral arterial disease
* Myocardial infarction or hospitalization within the previous 6 months
* Symptomatic orthostatic hypotension
* Hypertension in poor pharmacological control (diastolic> 95 mmHg, systolic> 160 mmHg)
* Significant neurological conditions that impair motor or cognitive function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
6 Minutes Walking Test | baseline,3 months,6 months
  The change in functional capacity calculated as the difference between the baseline 6 Minutes Walking Test assessment and the 3 and 6 month assessment measured with the G-Walk (BTS Bioengineering S.p.A).

SECONDARY OUTCOMES:
Functional Independence Score in Hemophilia (FISH) | baseline,3 months,6 months
  It is a questionnaire which is carried out by an operator to evaluate autonomy in carrying out eight activities of daily life: personal hygiene, eating, dressing, transferring from chairs, squatting, walking, climbing stairs, running. Each activity is measured according to the amount of assistance needed to perform it.
Hemophilia joint health score (HJHS) | baseline,3 months,6 months
  It is a scale compiled by an operator to evaluate the health status of the joints. The HJHS measures joint health in the domains of body structure and function (biomechanics) of the structures most frequently affected by hemorrhage in patients with hemophilia: the knees, ankles, and elbows.
Tampa Scale of Kinesiophobia - (TSK) | baseline,3 months,6 months
  It is a questionnaire filled in by the patient to assess fear of movement. This scale is an international evaluation parameter with which a persistent and constant, completely unjustified concern in carrying out movements for fear of causing pain or damage is highlighted.
Hemophilia Activity List (HAL) | baseline,3 months,6 months
  It is a questionnaire filled in by the patient on activity limitations. The HAL scale measures the impact of haemophilia on functional abilities in adults. It is made up of 42 questions investigating 7 domains: 1. Lying / Sitting / Kneeling / Standing, 2. Leg functions, 3. Arm functions, 4. Transport, 5. Personal care, 6. Household activities, 7. Leisure and sporting activities.
Balance - Single leg stand test | baseline,3 months,6 months
  The test should be performed with eyes open and hands on the hips. Instruct the patient to stand on one leg unassisted, starting when the patient's foot leaves the ground and stopping the time the patient's foot touches the ground and/or when their hands leave the hips. Abnormal values may indicate conditions such as peripheral neuropathy, intermittent claudication, or other conditions that may impair balance
Balance - Time Up and Go (TUG) | baseline,3 months,6 months
  The TUG is a general physical performance test used to assess mobility, balance and locomotor performance in people with potential balance disturbances. More specifically, it assesses the ability to perform sequential motor tasks relative to walking and turning.
Pain (VAS - Visual Analogue Scale ) | baseline,3 months,6 months
  Pain measured by VAS (Visual Analogue Scale) on target joint
Muscle strenght- 30" Chair stand test | baseline,3 months,6 months
  The purpose of this test in to evaluate leg strength and endurance, by counting the number of times the patient comes to a full standing position in 30 seconds
Muscle strenght-Arm curl test | baseline,3 months,6 months
  this test evaluates functional upper extremity fitness of adults, with the goal is to complete as many curls (through the entire available range of motion) in 30 seconds
Muscle strenght- Hand held measuring of hip and knee flexors/extensors | baseline,3 months,6 months
  Measure the muscle strenght of hip and knee flexors/extensors by using a Hand held

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Bo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iorio A, Stonebraker JS, Chambost H, Makris M, Coffin D, Herr C, Germini F; Data and Demographics Committee of the World Federation of Hemophilia. Establishing the Prevalence and Prevalence at Birth of Hemophilia in Males: A Meta-analytic Approach Using National Registries. Ann Intern Med. 2019 Oct 15;171(8):540-546. doi: 10.7326/M19-1208. Epub 2019 Sep 10. PMID 31499529
- [Background] Lee CA, Berntorp EE, Keith Hoots W; Textbook of Hemophilia 3th Edition 2014 Wiley Ed;
- [Background] Gurcay E, Eksioglu E, Ezer U, Cakir B, Cakci A. A prospective series of musculoskeletal system rehabilitation of arthropathic joints in young male hemophilic patients. Rheumatol Int. 2008 Apr;28(6):541-5. doi: 10.1007/s00296-007-0474-7. Epub 2007 Oct 18. PMID 17943258
- [Background] Hill K, Fearn M, Williams S, Mudge L, Walsh C, McCarthy P, Walsh M, Street A. Effectiveness of a balance training home exercise programme for adults with haemophilia: a pilot study. Haemophilia. 2010 Jan;16(1):162-9. doi: 10.1111/j.1365-2516.2009.02110.x. Epub 2009 Oct 5. PMID 19804383
- [Background] Srivastava A, Brewer AK, Mauser-Bunschoten EP, Key NS, Kitchen S, Llinas A, Ludlam CA, Mahlangu JN, Mulder K, Poon MC, Street A; Treatment Guidelines Working Group on Behalf of The World Federation Of Hemophilia. Guidelines for the management of hemophilia. Haemophilia. 2013 Jan;19(1):e1-47. doi: 10.1111/j.1365-2516.2012.02909.x. Epub 2012 Jul 6. PMID 22776238
- [Background] Nied RJ, Franklin B. Promoting and prescribing exercise for the elderly. Am Fam Physician. 2002 Feb 1;65(3):419-26. PMID 11858624
- [Background] Bennell KL, Hinman RS, Metcalf BR, Buchbinder R, McConnell J, McColl G, Green S, Crossley KM. Efficacy of physiotherapy management of knee joint osteoarthritis: a randomised, double blind, placebo controlled trial. Ann Rheum Dis. 2005 Jun;64(6):906-12. doi: 10.1136/ard.2004.026526. PMID 15897310
- [Background] Mulvany R, Zucker-Levin AR, Jeng M, Joyce C, Tuller J, Rose JM, Dugdale M. Effects of a 6-week, individualized, supervised exercise program for people with bleeding disorders and hemophilic arthritis. Phys Ther. 2010 Apr;90(4):509-26. doi: 10.2522/ptj.20080202. Epub 2010 Mar 4. PMID 20203091
- [Background] Gomis M, Querol F, Gallach JE, Gonzalez LM, Aznar JA. Exercise and sport in the treatment of haemophilic patients: a systematic review. Haemophilia. 2009 Jan;15(1):43-54. doi: 10.1111/j.1365-2516.2008.01867.x. Epub 2008 Aug 21. PMID 18721151
- [Background] Ettinger WH Jr, Burns R, Messier SP, Applegate W, Rejeski WJ, Morgan T, Shumaker S, Berry MJ, O'Toole M, Monu J, Craven T. A randomized trial comparing aerobic exercise and resistance exercise with a health education program in older adults with knee osteoarthritis. The Fitness Arthritis and Seniors Trial (FAST). JAMA. 1997 Jan 1;277(1):25-31. PMID 8980206
- [Background] Roddy E, Zhang W, Doherty M. Aerobic walking or strengthening exercise for osteoarthritis of the knee? A systematic review. Ann Rheum Dis. 2005 Apr;64(4):544-8. doi: 10.1136/ard.2004.028746. PMID 15769914
- [Background] Fransen M, McConnell S, Bell M. Therapeutic exercise for people with osteoarthritis of the hip or knee. A systematic review. J Rheumatol. 2002 Aug;29(8):1737-45. PMID 12180738
- [Background] Fransen M, McConnell S, Hernandez-Molina G, Reichenbach S. Exercise for osteoarthritis of the hip. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007912. doi: 10.1002/14651858.CD007912. PMID 19588445
- [Background] World Federation Guidelines of Hemophilia - 2nd Edition
- [Background] Siqueira TC, Dominski FH, Andrade A. Effects of exercise in people with haemophilia: An umbrella review of systematic reviews and meta-analyses. Haemophilia. 2019 Nov;25(6):928-937. doi: 10.1111/hae.13868. Epub 2019 Oct 30. PMID 31667968
- [Background] Deniz V, Guzel NA, Lobet S, Antmen AB, Sasmaz HI, Kilci A, Boyraz OC, Gunasti O, Kurdak SS. Effects of a supervised therapeutic exercise program on musculoskeletal health and gait in patients with haemophilia: A pilot study. Haemophilia. 2022 Jan;28(1):166-175. doi: 10.1111/hae.14444. Epub 2021 Oct 22. PMID 34687122
- [Background] Poonnoose PM, Manigandan C, Thomas R, Shyamkumar NK, Kavitha ML, Bhattacharji S, Srivastava A. Functional Independence Score in Haemophilia: a new performance-based instrument to measure disability. Haemophilia. 2005 Nov;11(6):598-602. doi: 10.1111/j.1365-2516.2005.01142.x. PMID 16236109
- [Background] Ribeiro T, Abad A, Feldman BM. Developing a new scoring scheme for the Hemophilia Joint Health Score 2.1. Res Pract Thromb Haemost. 2019 May 20;3(3):405-411. doi: 10.1002/rth2.12212. eCollection 2019 Jul. PMID 31294328
- [Background] Monticone M, Giorgi I, Baiardi P, Barbieri M, Rocca B, Bonezzi C. Development of the Italian version of the Tampa Scale of Kinesiophobia (TSK-I): cross-cultural adaptation, factor analysis, reliability, and validity. Spine (Phila Pa 1976). 2010 May 20;35(12):1241-6. doi: 10.1097/BRS.0b013e3181bfcbf6. PMID 20216338
- [Background] van Genderen FR, Westers P, Heijnen L, de Kleijn P, van den Berg HM, Helders PJ, van Meeteren NL. Measuring patients' perceptions on their functional abilities: validation of the Haemophilia Activities List. Haemophilia. 2006 Jan;12(1):36-46. doi: 10.1111/j.1365-2516.2006.01186.x. PMID 16409173
- [Background] Benton MJ, Alexander JL. Validation of functional fitness tests as surrogates for strength measurement in frail, older adults with chronic obstructive pulmonary disease. Am J Phys Med Rehabil. 2009 Jul;88(7):579-83; quiz 584-6, 590. doi: 10.1097/PHM.0b013e3181aa2ff8. PMID 19542782
- [Background] Hebert LJ, Maltais DB, Lepage C, Saulnier J, Crete M, Perron M. Isometric muscle strength in youth assessed by hand-held dynamometry: a feasibility, reliability, and validity study. Pediatr Phys Ther. 2011 Fall;23(3):289-99. doi: 10.1097/PEP.0b013e318227ccff. PMID 21829128
- [Background] Hunt MA, McManus FJ, Hinman RS, Bennell KL. Predictors of single-leg standing balance in individuals with medial knee osteoarthritis. Arthritis Care Res (Hoboken). 2010 Apr;62(4):496-500. doi: 10.1002/acr.20046. PMID 20391504
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Louangrath, Paul. (2018). Reliability and Validity of Survey Scales. 10.5281/zenodo.1322695.
- [Background] World Health Organization. Global action plan on physical activity 2018-2030: more active people for a healthier world. 2018. http://apps.who.int/iris/bitstream/handle/10665/272722/9789241514187-eng.pdf

DOCUMENTS (1):
  • Study Protocol (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT06580340/Prot_000.pdf